CLINICAL TRIAL: NCT03936218
Title: A Two Arm, Multi Centric, Randomised, Open Label, Parallel Study to Compare Pharmacodynamics of Subcutaneous Goserelin 10.8mg Injection (Sponsor) With ZOLADEX® 10.8mg Injection (AstraZeneca) in Patients With Advanced Prostate Cancer
Brief Title: Goserelin 10.8mg Injection in Treatment of Advanced Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF 161
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-05

CONDITIONS: Advanced Prostate Cancer
MeSH Terms: interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inj. Goserelin (Test) Subcutaneously (Experimental): 10.8 mg, Subcutaneously at every 3 month
  Interventions: Drug: Inj. Goserelin (Test) Subcutaneously
- Inj. Zoladex (Reference) Subcutaneously (Active Comparator): 10.8 mg, Subcutaneously at every 3 month
  Interventions: Drug: Inj. Zoladex (Reference) Subcutaneously

INTERVENTIONS:
Drug: Inj. Goserelin (Test) Subcutaneously — 10.8 mg, subcutaneously at every 3 month
  Other Names: Goserelin
  Arms: Inj. Goserelin (Test) Subcutaneously
Drug: Inj. Zoladex (Reference) Subcutaneously — 10.8 mg, Subcutaneously at every 3 month
  Other Names: Zoladex
  Arms: Inj. Zoladex (Reference) Subcutaneously

SUMMARY:
A two arm, multi centric, randomized, open label, parallel, two doses pharmacodynamics study in patients with advanced prostate cancer.

DETAILED DESCRIPTION:
A phase III, two arm, multi centric, randomized, open label, parallel, two doses pharmacodynamics study in patients with advanced prostate cancer. Each patient will have 25 visits total. Total duration of the study will be 183 days (including up to 14 days of screening).

ELIGIBILITY:
Inclusion Criteria:

1. Male patient with age of 18 to 75 years (Both inclusive)
2. Body mass index (BMI) between 18.5 and 30 kg/m². (Both inclusive)
3. Patient with a confirmed advanced prostatic adenocarcinoma. (TNM stage III or IV or recurrent metastatic disease) who are scheduled to start Goserelin therapy as per Investigator discretion. Note: Stage III (T1-T2, N0, M0, PSA level is 20 or more, Grade Group 1-4 or T3--T4, N0, M0, any PSA, Grade Group 1-4 or any T, N0, M0, any PSA, Grade Group 5). Stage IV (any T, N1, M0, any PSA, any Grade Group or any T, N0, M1, any PSA, any Grade Group)
4. Serum testosterone level >2.5 ng/mL for age of 20 to 49 (both inclusive) and >1.9 ng/mL for age ≥ 50 at screening. (Screening sample for Serum testosterone level should be taken before 10:00 am in the morning).
5. Patient must be able to give informed consent for participation in the trial.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
7. Adequate bone marrow function, renal function, liver function.
8. Patient should have recovered from any toxic effects of previous chemotherapy as judged by the Investigator.
9. Patients with life expectancy of at least 1 year as judged by the Investigator.
10. Patient or his partner willing to use an effective method as mentioned below of contraception during the study:

    * Tubal sterilization (tubal ligation performed more than one month before Study Day 1; transcervical tubal occlusion procedure performed more than six months before Study Day 1)
    * Barrier method (cervical cap, diaphragm, contraceptive sponge, vaginal spermicide, female condom, or male condom)
    * Two barrier methods used together (cervical cap, diaphragm, contraceptive sponge, or vaginal spermicide plus a male or female condom) Absolute sexual abstinence (no sexual intercourse or genital contact with a female partner). If the patient becomes sexually active during the study, then he is required to use a double barrier method of contraception.

Exclusion Criteria:

1. Evidence of severe urinary tract obstruction with anticipated urinary retention, in the opinion of the Investigator, taking into account medical history, clinical observations and symptoms.
2. Patients who are scheduled to receive any chemotherapy/radiotherapy in addition to goserelin.
3. Patients who are already on GnRH receptor agonist or antagonist therapy directed for prostate cancer.
4. Patients who have previously failed on GnRH receptor agonist or antagonist therapy for prostate cancer.
5. Presence of life-threatening metastatic visceral disease, defined as extensive hepatic involvement, or any degree (proven or suspected) of brain or leptomeningeal involvement (past or present) or symptomatic pulmonary lymhangitic spread. Patients with discrete pulmonary parenchymal metastases are eligible, provided their respiratory function is not compromised as a result of disease.
6. Patients who are intended to be started on any medication apart from study drug that can have impact on any of the study endpoints.
7. Patients with spinal cord compression (in the opinion of the Investigator), taking into account medical history, clinical observations and symptoms.
8. Excruciating, severe bone pain which is due to extensive metastatic osseous deposits.
9. Patient has "currently active" second malignancy, other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy if they have completed therapy >5 years previously and have no known evidence of residual or recurrent disease.
10. Patients with confirmed signs or symptoms related to cerebral metastasis or radiographically confirmed brain metastasis.
11. Patients with a clinically significant medical condition other than advanced prostate cancer including but not limited to renal, hepatic, gastrointestinal, endocrine, cardiovascular, neurological or psychiatric disease, alcohol or substance abuse, or any other condition that may affect the patient's health or the outcome of the trial as judged by the investigator.
12. Patients with a known hypersensitivity to GnRH, GnRH-agonist analogues or any of the components in IMP.
13. History of orchiectomy, adrenalectomy or hypophysectomy.
14. Patients receiving anticoagulation medications.
15. Patients with uncontrolled diabetes mellitus (HbA1c > 8 % as per ADA) at randomization (those who have controlled blood sugar (fasting) will be eligible for randomization)
16. Uncontrolled hypertension (systolic blood pressure [BP] >140 or diastolic BP >90mm Hg) or uncontrolled cardiac arrhythmias. (Patients with hypertension controlled by antihypertensive therapies are eligible).
17. Patients with a QTc>450ms on the ECG at screening.
18. History of clinically significant cardiovascular disorder.
19. Use of any recreational drugs (cocaine, amphetamines, barbiturates, benzodiazepines, cannabinoids and morphine) or history of drug or alcohol abuse within the past 1 year, as judged by the Investigator, or a positive result on the urine drug/alcohol screen which is not consistent with current medical treatment.
20. Concomitant use of medicinal products known to prolong the QT interval or medicinal products able to induce Torsade de pointes such as class IA (e.g. quinidine, disopyramide) or class III (e.g. amiodarone, sotalol, dofetilide, ibutilide) antiarrhythmic medicinal products, methadone, moxifloxacin, antipsychotics.
21. A positive hepatitis screen including hepatitis B surface antigen or HCV antibodies.
22. Patients who test positive for HIV and/or syphilis.
23. The receipt of an investigational product, or participation in a drug research study within a period of 30 days prior screening or 5 half-lives within the last dose of investigational product, whichever is longer. Current use of any drugs that are known to interfere with goserelin metabolism or to cause a drug-drug interaction.
24. Donation / loss of blood/plasma or blood product (without replenishment) (1 unit or 350 mL) within 180 days prior to receiving the first dose of study medicine.
25. Patients with a mental incapacity, unwillingness, or language barrier that precludes the ability to understand or cooperate with study procedures.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
To evaluate and compare the pharmacodynamics of test product against reference product and establish non inferiority. | 24 weeks
  Proportion of patients achieving castrate level of serum testosterone (Serum testosterone ≤ 0.5 ng/ml) at the end of 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mahatma Gandhi Cancer Hospital & Research Institute, Visakhapatnam, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.